CLINICAL TRIAL: NCT05159050
Title: Phase I Trial of Intraperitoneal Paclitaxel-loaded Tumor Penetrating Microparticles (TPM) for Treatment of Peritoneal Carcinomatosis
Brief Title: Intraperitoneal Paclitaxel-loaded TPM for Treatment of Peritoneal Carcinomatosis
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Drug supply issues
Sponsor: Carlos Chan (Other)
Collaborators: Institute of Quantitative Systems Pharmacology (IQSP) (Unknown)
Responsible Party: Sponsor-Investigator, Carlos Chan, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202105008
Record Dates: First submitted 2021-11-08; First posted 2021-12-15 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Peritoneal Carcinomatosis
MeSH Terms: conditions — Peritoneal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intraperitoneal paclitaxel-loaded tumor penetrating microparticles (TPM) (Experimental): Paclitaxel-loaded tumor penetrating microparticles (TPM), dose escalation starting at 50 mg/m^2 instilled in the peritoneal cavity at study start and again 6-8 weeks after the first TPM treatment.
  Interventions: Drug: Paclitaxel-loaded tumor penetrating microparticles

INTERVENTIONS:
Drug: Paclitaxel-loaded tumor penetrating microparticles — Paclitaxel-loaded TPM, suspended in 0.5 L of 0.1% (w/v) polysorbate 80 in 0.9% sodium chloride is instilled into the peritoneal cavity over 3 to 5 minutes. Mixing of TPM is achieved by putting patient in 5 different positions for about 80 minutes.
  Dose escalation, the starting dose of TPM is 50 mg/m^2 paclitaxel-equivalents. Dose escalation will follow the Accelerated Titration Design. The dose levels to which patients will be assigned in sequential cohorts are listed below.
  Dose escalation schedule of TPM, Dose Level 1*: 50 mg/m^2; Dose Level 2: 100 mg/m^2; Dose Level 3: 135 mg/m^2; Dose Level 4: 175 mg/m^2; Dose Level 5: 200 mg/m^2
  *Starting Dose

SUMMARY:
A first-in-human, unblinded, phase I trial of Paclitaxel-loaded tumor penetrating microparticles (TPM) in peritoneal carcinomatosis patients who are not eligible for standard-of-care therapeutic interventions.

DETAILED DESCRIPTION:
This is a first in human study of Paclitaxel-loaded TPM, suspended in 0.5 L of 0.1% polysorbate 80 in normal saline instilled into the peritoneal cavity.

An enrolled patient will (a) undergo laparoscopy during which time the hydrostatic pressures at different locations within the peritoneal cavity are measured, pretreatment tumors are biopsied and peritoneal catheter is placed, (b) receive intraperitoneal TPM during index hospital stay, and (c) followed-up to evaluate treatment-related toxicity and response. The pharmacokinetics of TPM and paclitaxel in peritoneal fluid and systemic blood samples will be measured. Second dose of TPM is given in clinic if no disease progression or significant AEs.

This is a dose escalation study. Dose escalation will proceed using an accelerated titration design (ATD) with intra-patient dose escalation.

In the event either:

* 1 patient exhibits DLT during the first course of treatment or
* 2 patients exhibit grade 2 study drug-related (attribution of probable or definite) toxicity during the first course of treatment.

The design switches to a standard 3+3 design at the dose that triggered the switch-two additional patients are accrued at this dose level. Decisions on when and how to escalate if the design switches to a 3+3 are described in the protocol section 6.3

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document
* Have pathology proven peritoneal carcinomatosis (PC) due to colorectal, ovarian, gastric, pancreatic, appendiceal cancer or mesothelioma, or suspected peritoneal metastasis based on radiological findings. (Patient to come off study if no pathology evidence of peritoneal metastasis at the time of surgery)
* No other standard treatment options are available
* Measurable intraperitoneal disease by RECIST v1.1 criteria , or by radiological PCI scoring when RECIST is not feasible, on imaging studies
* 18 to 75 years of age
* Have an ECOG performance of 0 to 2
* Have adequate organ and bone marrow functions as indicated by:
* Leukocytes ≥ 3000/mcL
* Absolute neutrophil count ≥ 1500/mcL
* Platelets ≥ 100000/mcL
* Total bilirubin within normal institutional limits
* AST (SGOT) < 3 x institutional upper limit of normal
* ALT (SPGT) < 3 x institutional upper limit of normal
* Medically fit for surgery. Defined as: Patients who are able to undergo general anesthesia for abdominal surgery and have a metabolic equivalent (METs) ≥ 4
* Have adequate contraception, as follows:

  1. Women of child-bearing potential and men with partners of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 10 months beyond the last dose of TPM. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
  2. A woman of child-bearing potential is any female (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
* has not undergone a hysterectomy or bilateral oophorectomy; or
* has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)

  c. Men with partners of child bearing potential must use barrier contraceptive

  d. Men of child-bearing potential must not donate sperm while on this study and for 7 months after the last dose of TPM

Acceptable forms of birth control are listed below:

* One Barrier method (cervical cap with spermicide plus male condom; diaphragm with spermicide plus male condom) OR
* Hormonal method (oral contraceptives, implants, or injections) or an intrauterine device (e.g., Copper-T)

Exclusion Criteria:

* Presence of mucinous ascites
* Evidence of extra-peritoneal metastases
* Current or expected use of other investigational agents
* Received systemic chemotherapy or radiotherapy within 3 weeks prior to study enrollment or not recovering from adverse events (e.g., recovery to ≤ Grade 1)
* Abdominal cavity deemed not accessible by treating surgeon due to prior abdominal surgery
* History of allergic reactions to paclitaxel, PLG co-polymer, mannitol, or polysorbate 80
* Uncontrolled intercurrent illness
* Currently active second malignancy other than non-melanoma skin cancer
* Pregnancy, nursing, or plans to become pregnant for the duration of study participation including 10 months beyond the last dose of TPM
* Grade 2 or higher peripheral neuropathy
* CrCL ≤ 4 mL/min
* Actively treated for other malignancy
* Patients with HIV or Hepatitis B/C requiring the use of ART agents

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2026-01-14 (Estimated); Study Completion 2026-01-14 (Estimated)

PRIMARY OUTCOMES:
Assess safety of intraperitoneal Paclitaxel-loaded Tumor Penetrating Microparticles (TPM) | 12 Weeks
  The incidence of treatment-emergent adverse events will be summarized by system organ class and/or preferred term, type of adverse event, severity (based on NCI CTCAE v5.0 grades), and relation to study treatment using the safety population.
Determine the maximum tolerated dose (MTD) of intraperitoneal Paclitaxel-loaded Tumor Penetrating Microparticles (TPM) | 4 Weeks
  Dose escalation will proceed using an accelerated titration design (ATD). Subjects will be observed for 4 weeks after the first course of TPM treatment for any potential dose limiting toxicities (DLT). The MTD is defined as the highest dose level for which at most 1 out of 6 patients experience a DLT.

SECONDARY OUTCOMES:
Assess potential therapeutic efficacy of intraperitoneal Paclitaxel-loaded Tumor Penetrating Microparticles (TPM) | 12 Weeks
  Tumor response will be measured by RECIST v1.1 to determine potential effective doses of intraperitoneal Paclitaxel-loaded TPM.
Measure area-under-drug concentration-time curve of Paclitaxel and tumor penetrating microparticles (TPM) in blood and peritoneal fluid | 8 Weeks
  Paclitaxel-loaded TPM pharmacokinetics will be described using summary statistics, such as mean and range, and graphical displays.
Measure maximum drug concentration of Paclitaxel and tumor penetrating microparticles (TPM) in blood and peritoneal fluid | 8 Weeks
  Paclitaxel-loaded TPM pharmacokinetics will be described using summary statistics, such as mean and range, and graphical displays.
Assess whether Paclitaxel-loaded Tumor Penetrating Microparticles (TPM) induce immune response in the peritoneal cavity | 8 Weeks
  The presence or absence of T cell infiltration in peritoneal cavity.
Assess whether intra-abdominal pressure is location-dependent | Day 1 on study
  Intra-abdominal hydrostatic pressures at various intraperitoneal locations will be measured at the time of laparoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Chan, MD, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals & Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No